CLINICAL TRIAL: NCT07257406
Title: The Use of Intravenous Dexamethasone for Post-operative Pain After Cesarean Delivery Under Neuraxial Anesthesia.
Brief Title: Dexamethasone for Post-operative Pain After Cesarean Delivery Under Neuraxial Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valerie Zaphiratos (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, Valerie Zaphiratos, Associate Professor of Anesthesiology, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-1840
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Cesarean Delivery; Dexamethasone
Keywords: pregnancy; dexamethasone; cesarean; pain
MeSH Terms: conditions — Pain | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone (IV)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone (IV) — Dexamethasone 8 mg IV will be given 5 minutes after cord clamping in the interventional arm.
  Arms: Dexamethasone
Drug: Placebo — This arm will receive 2 ml of saline 5 min after cord clamping.
  Arms: Placebo

SUMMARY:
After surgery pain in women who have had a cesarean delivery is a determining factor in the quality and duration of their hospital stay. Insufficient pain relief can lead to longer hospitalization and long term pain, which can result in long term use of pain medication. A classic method to alleviate pain after cesarean delivery is by injecting morphine into the spinal fluid, in the women's back, in addition to prescribing morphine by mouth as needed after the surgery. However, the negative effects associated with morphine and morphine-like drugs, limit the doses used, their pain relief capacity, and can negatively affect the after surgical experience of women. An approach which uses pain relief that acts on different pain pathways to treat after surgery pain helps limit the negative effects of different drugs. The potential benefit of dexamethasone as pain relief in women who have had a cesarean delivery is all the more interesting because of its minimal negative effects compared to morphine-like drugs. Its low cost, its effectiveness to prevent nausea, and its impact on the general condition of patients make dexamethasone even more attractive.

DETAILED DESCRIPTION:
Postoperative pain in patients who have undergone a cesarean delivery is a determining factor in the quality and duration of their hospital stay. Suboptimal analgesia can lead to prolonged hospitalization and chronic pain, which can result in chronic use of pain medication. Treatment of post-operative pain after cesarean delivery uses intrathecal morphine, and the use of opioids as needed post-operatively. However, the side effects associated with opioids limit the doses used, their analgesic efficacy, and adversely affect the postoperative experience of patients. The multimodal approach to postoperative pain allows for analgesia that acts on different pain mechanisms while limiting the adverse effects of different drugs. The potential benefits of dexamethasone as a co-analgesic in women who have had a cesarean section are all the more interesting because of its minimal adverse effects compared to opioids. Its low cost, its effectiveness as antiemetic prophylaxis, and its impact on the general condition of patients make dexamethasone even more attractive.

In this randomised controlled trial, 100 patients are to be recruited and randomised to one of two groups. Both groups will receive standard treatment. In addition to standard treatment, the first group will receive dexamethasone 8 mg IV after umbilical cord clamping and the other group will receive a placebo.

The patients will be followed for 24 hours post-operatively. Their pain levels at rest and during movement will be recorded on an 11 point pain scale. The dose of hydromorphone used in the first 24 hours will be recorded. The patients are also asked to complete the QOR-40 questionnaire, which aims to assess the quality of their postoperative recovery. The primary outcome is the pain on an 11 point scale at the first rise 6 hours post-operatively.

The investigators hypothesize that dexamethasone will improve pain scores and diminish opioid use in the first 24 hours post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Cesarean delivery
* Planned spinal or combined neuraxial anesthesia
* Presence of an investigator in the delivery room
* Pregnancy > 34 weeks gestation

Exclusion Criteria:

* Cesarean delivery under general anesthesia
* Inability to understand French or English
* Allergy or hypersensitivity to dexamethasone
* Allergy to hydromorphone
* Allergy to NSAIDs
* Acute kidney injury or chronic kidney failure
* Preeclampsia
* Extremely urgent cesarean section
* Urgent cesarean section with non-reassuring fetal monitoring
* Known maternal heart disease
* High-grade placental abnormality
* Diabetes (pregnancy or pre-existing)
* Systemic infection, sepsis, fever
* Regular use of dexamethasone in the last year
* Weight greater than 120 kg and less than 70 kg
* Height less than 150 cm
* Chronic pain and/or chronic use of opioids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Score (VAS) 6 hours post-operatively at first rise | 6 hours post-operatively
  Visual Analog Pain Score (VAS), from 0 to 10, when patients first stand out of bed 6 hours post-operatively. A score of 0 on 10 being no pain, and a score of 10 on 10 being the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
If a researcher needs IPD for a meta-analysis for instance, they can contact me.

REFERENCES:
- [Background] Mohtadi A, Nesioonpour S, Salari A, Akhondzadeh R, Masood Rad B, Aslani SM. The effect of single-dose administration of dexamethasone on postoperative pain in patients undergoing laparoscopic cholecystectomy. Anesth Pain Med. 2014 Aug 13;4(3):e17872. doi: 10.5812/aapm.17872. eCollection 2014 Aug. PMID 25237639
- [Background] Shahraki AD, Feizi A, Jabalameli M, Nouri S. The effect of intravenous Dexamethasone on post-cesarean section pain and vital signs: A double-blind randomized clinical trial. J Res Pharm Pract. 2013 Jul;2(3):99-104. doi: 10.4103/2279-042X.122370. PMID 24991614
- [Background] Cardoso MM, Leite AO, Santos EA, Gozzani JL, Mathias LA. Effect of dexamethasone on prevention of postoperative nausea, vomiting and pain after caesarean section: a randomised, placebo-controlled, double-blind trial. Eur J Anaesthesiol. 2013 Mar;30(3):102-5. doi: 10.1097/EJA.0b013e328356676b. PMID 23022704